CLINICAL TRIAL: NCT03222310
Title: Effect of a Potent CYP3A and P-gp Inhibitor (Itraconazole) on Ipatasertib Pharmacokinetics in Healthy Subjects
Brief Title: A Study to Evaluate the Effect of a Potent Cytochrome P450 (CYP) 3A Inhibitor on Ipatasertib
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GP30057
Record Dates: First submitted 2017-07-17; First posted 2017-07-19 (Actual); Last update posted 2017-11-09 (Actual); Status verified 2017-11

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — ipatasertib; Itraconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Ipatasertib (Experimental): Participants will receive one 100 milligram (mg) ipatasertib tablet orally on Day 1 of treatment in treatment period 1 followed by two 100 mg itraconazole capsules orally on Days 15 to 23 along with one 100 mg of ipatasertib on Day 19 in treatment period 2. Both the treatment period will be separated by a washout period of 14 days.
  Interventions: Drug: Ipatasertib; Drug: Itraconazole

INTERVENTIONS:
Drug: Ipatasertib — Ipatasertib 100 mg tablet orally once daily.
Drug: Itraconazole — Itraconazole 100 mg capsules orally once daily.

SUMMARY:
This study will be a single center, open-label, 2-period, fixed-sequence, Phase 1 drug-drug interaction study in healthy subjects. The primary purpose of this study is to evaluate the effect of itraconazole on the PK of ipatasertib and its primary metabolite (G-037720).

ELIGIBILITY:
Inclusion Criteria:

* Within body mass index (BMI) range 18.5 to 32.0 kg/m2, inclusive
* In good health, determined by no clinically significant findings from medical history, 12-lead ECG, and vital signs
* Clinical laboratory evaluations (including chemistry panel [fasted at least 8 hours], hematology, and urinalysis [UA] with complete microscopic analysis within the reference range for the test laboratory, unless deemed not clinically significant by the Investigator)
* Negative test for selected drugs of abuse at Screening (does not include alcohol) and at Check-in (Day -2)
* Negative hepatitis panel (hepatitis B surface antigen and hepatitis C virus antibody) and negative human immunodeficiency virus (HIV) antibody screens

Exclusion Criteria:

* Significant history or clinical manifestation of any metabolic, allergic, dermatological, hepatic, renal, hematological, pulmonary, cardiovascular, GI, neurological, or psychiatric disorder (as determined by the Investigator)
* History of diabetes requiring insulin or fasting glucose ≥160 mg/dL
* History of significant hypersensitivity, intolerance, or allergy to any drug compound, food, or other substance, unless approved by the Investigator
* history of stomach or intestinal surgery or resection, or other GI disorder that would potentially alter absorption and/or excretion of orally administered drugs, except that appendectomy, hernia repair, and/or cholecystectomy will be allowed
* history or presence of an abnormal ECG, which, in the Investigator's opinion, is clinically significant

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2017-07-18 (Actual); Primary Completion 2017-09-06 (Actual); Study Completion 2017-09-06 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) of ipatasertib and its Metabolite (G-037720) | Pre-dose, 0.167, 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 36, 48, 72, 96, 120, 144 hours post dose on Day 1 and 19; 168, 192 hours post dose on Day 19
  Cmax is the maximum observed concentration.
Area Under the Plasma Concentration-Time Curve From Time Zero to Extrapolated Infinite Time (AUC[0-inf]) of Ipatasertib and its Metabolite (G-037720) | Pre-dose, 0.167, 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 36, 48, 72, 96, 120, 144 hours post dose on Day 1 and 19; 168, 192 hours post dose on Day 19
  AUC(0-inf) is the area under the plasma concentration versus time curve (AUC) from time zero (pre-dose) to extrapolated infinite time (0-inf). AUC is a measure of the plasma concentration of a drug over time.
Area Under the Plasma Concentration-Time Curve From Hour 0 to the Last Measureable Concentration (AUC0-t) of Ipatasertib and its Metabolite (G-037720) | Pre-dose, 0.167, 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 36, 48, 72, 96, 120, 144 hours post dose on Day 1 and 19; 168, 192 hours post dose on Day 19
  Area Under the Plasma Concentration-Time Curve From Hour 0 to the Last Measureable Concentration (AUC0-t) will be reported.

SECONDARY OUTCOMES:
Number of Participants Who Experienced at Least 1 Adverse Event | Up to 28 days after the last dose of the study drug (approximately up to 51 days)
  An adverse event is any untoward medical occurrence in a patient administered a pharmaceutical product and which does not necessarily have to have a causal relationship with the treatment. An adverse event can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a pharmaceutical product, whether or not considered related to the pharmaceutical product. Preexisting conditions which worsen during a study are also considered as adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (1):
- Covance Research Unit - Dallas, Dallas, Texas, United States